CLINICAL TRIAL: NCT06423651
Title: Benefits of Combining Metacognitive Training (MCT) With Cognitive Remediation (CR) in the Recovery of Patients With Psychotic Spectrum Disorders (CR+MCTp)
Brief Title: Benefits of Combining MCT With CR in the Recovery of Patients With Psychotic Spectrum Disorders
Acronym: CR+MCTp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Autonoma de Barcelona (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Consorci Sanitari de Terrassa (Other); Hospital de Mataró (Other); Centre d'Higiene Mental Les Corts (Other); Fundació Els 3 Turons (Unknown); Hospital San Carlos, Madrid (Other); Andaluz Health Service (Other Government); Institut d'Assistència Sanitària (Other); Ministerio de Ciencia, Innovación y Universidades (Unknown); Hospital Son Espases (Other); Parc Taulí Hospital Universitari (Other); Servicio Cántabro de Salud (Other)
Responsible Party: Principal Investigator, Ana Barajas Velez, Associate Professor, Universitat Autonoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PID2020-118907RA-I00
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Delusional Disorder; Brief Psychotic Disorder; Schizoaffective Disorder; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Metacognitive Training; MCT; Cognitive Remediation; Psychotic disorder; Psychosis; Cognitive functions; Cognitive biases; Neurocognitive improvement
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: This will be a randomized clinical trial in which one group will receive combined REHACOP + MCT therapy and another group will receive therapy with MCT alone. The metacognitive treatment will have the same characteristics in the two treatment conditions. Randomisation of the patients for receiving one of the two treatments will be carried out using a random number list based on the order of access to their reference centre. The evaluator will be blinded to the treatment group to which the patient assessed belongs.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REHACOP+MCT therapy (Experimental): The participants will receive a combined therapy: Metacognitive Training (MCT) with Cognitive Remediation (CR).
  Interventions: Behavioral: Cognitive Remediation (REHACOP); Behavioral: Metacognitive Training (MCT)
- MCT alone (Active Comparator): The participants will receive Metacognitive Training (MCT)
  Interventions: Behavioral: Metacognitive Training (MCT)

INTERVENTIONS:
Behavioral: Cognitive Remediation (REHACOP) — REHACOP is a structured neuropsychological rehabilitation program that covers most of the cognitive deficits present in psychotic disorder: attention, learning and memory, executive functions, language, social cognition, daily life activities, social skills and psychoeducation. The modules of language, social cognition and psychoeducation will not be used in the present clinical trial. Each module includes a hierarchy of exercises based on the cognitive subarea to be worked on and the grade of difficulty demanded for the performance of each task.The format of the sessions will be the same as MCT, that is, groups of 6-10 patients who will receive weekly sessions of 45-60 minutes in length. In this case, the duration of the intervention will be 12 sessions.
  Arms: REHACOP+MCT therapy
Behavioral: Metacognitive Training (MCT) — The MCT consists in 8 weekly sessions of 45-60 minutes in length. Each group of patients should be made up of 6-10 patients. The material of the training program is available online at: http://www.uke.de/mkt. The material contains 16 powerpoint presentations (2 per each module), one manual and 6 pamphlets of tasks to do at home. The modules are as follows: Module 1: Attribution; Module 2: Jumping to conclusions (1st part); Module 3: Changing beliefs; Module 4: To emphatise (1st part); Module 5: Memory; Module 6: To emphatise (2nd part); Module 7: Jumping to conclusions (2nd part); and Module 8: Self-esteem and mood.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of combined REHACOP + MCT alone in persons with nonaffective psychotic disorder in terms of recovery. The main questions it aims to answer are:

* Does combined REHACOP + MCT therapy increase the clinical recovery in persons with nonaffective psychotic disorder (compared to MCT alone)?
* What is the impact of combined REHACOP + MCT therapy compared to MCT therapy alone on personal/psychological recovery, cognitive biases, and social cognition, taking gender differences into account?
* What is the durability of the effects of combined REHACOP + MCT therapy compared to MCT therapy alone on clinical recovery, personal recovery, cognitive biases, and social cognition in the long term?

Researchers will compare REHACOP+MCT therapy to MCT alone to see if there are differences in personal/psychological recovery.

Participants will:

* Participate in Metacognitive Training or in combined REHACOP + Metacognitive training therapy.
* Do 8 weekly sessions of 45-60 minutes (MCT group).
* Do 12 weekly sessions of 45-60 minutes (RECHACOP+MCT group).
* Visit the clinic for checkups and tests.
* Answer self-administered tests.

DETAILED DESCRIPTION:
This project is aimed at responding to one of the Challenges of the Spanish Strategy for Science, Technology and Innovation, specifically Challenge 1: Health, demographic change and well-being. One of the work areas that are located within this challenge is the Clinical and Translational Research based on the evidence of scientific and technological knowledge.The present proposal is clearly within the framework of clinical-translational investigation, since most of the entities participating attend persons with psychotic disorders, thereby ensuring the translation of investigation to the clinical setting. In addition, this project includes investigators with wide experience in psychological interventions in the target population and with previous experience in investigation in this area. Lastly, it is of note that the benefits of this investigation are not only of a scientific nature but also involve clinical investigation with a direct repercussion on improvement in the health care of people with psychotic disorders, enabling the design of new strategies of psychological interventions. Besides, the present proposal is aimed at responding to the challenges of our society, contributing to covering the needs of persons with psychotic disorder as well as developing the most effective therapeutic strategies to improve aspects related to clinical and personal recovery. Specifically, this project will allow making changes that will improve the quality of health care to the target population incorporating the combinated use of scientifically proven therapeutic strategies to health care services. In short, this project aims to promote innovation in the provision of mental health services, being the starting point in analyzing the efficacy of combined psychological therapies versus monotherapies address to improve of metacognitive processes.

- General and specific objectives. General objective: Compare the efficacy of combined REHACOP + MCT therapy vs. MCT alone in persons with nonaffective psychotic disorder in terms of recovery.

Specific objectives:

* Evaluate the effects of combined REHACOP + MCT therapy vs. MCT alone on clinical recovery (clinical remission and functional recovery, the latter understood in terms of cognitive, occupational and social functioning).
* Evaluate the effects of combined REHACOP + MCT therapy vs. MCT alone on personal/psychological recovery.
* Evaluate the effects of combined REHACOP + MCT therapy vs. MCT alone on cognitive biases and social cognition.
* Evaluate the effects of combined REHACOP + MCT therapy vs. MCT alone according to gender.
* Evaluate the effects of combined REHACOP + MCT therapy vs. MCT alone according to self-esteem, quality of life and stigma.
* Evaluate the maintenance of the effects of combined REHACOP + MCT therapy vs. MCT alone on clinical recovery, personal recovery, cognitive biases and social cognition in the long term.
* Methodology

Design:

This will be a randomised clinical trial in which one group will receive combined REHACOP + MCT therapy and another group will receive therapy with MCT alone. The metacognitive treatment will have the same characteristics in the two treatment conditions. Randomisation of the patients for receiving one of the two treatments will be carried out using a random number list based on the order of access to their reference centre. The evaluator will be blinded to the treatment group to which the patient assessed belongs.

Study subjects: The sample will be made up of people with non-affective psychotic disorder who are attended in any of the centres participating in the study which belong to the following entities:Consorci Sanitari de Terrassa; Hospital de Mataró; Instituto de Investigación Biomédica de Gerona (IdIBG); Parc Sanitari Sant Joan de Déu; Asociación Centro de Higiene Mental Les Corts; Hospital Sierrallana-Tres Mares; and UGC Salud Mental de Jaén.

Sample size: Considering that the investigators have no preliminary data on our principal objective in relation to clinical and personal recovery, the score obtained in the global assessment of functioning (GAF) at follow-up will be taken as a measure of outcome, since it is implicated in both clinical and functional recovery. The investigators used the data published in the article by Ochoa et al. (2017) in order to calculate the required sample size for this study. In this article, a difference of means of 5.73 points (SD=11.51) is obtained in the GAF scale from baseline and the follow-up at 6 months after the intervention. With these data, the necessary sample size has been estimated with an alpha of 0.05 and a power of 0.8. Taking into account 20% of possible losses to follow-up, the sample size has been calculated as 160 cases, 80 in each experimental arm (REHACOP + MCT vs. MCT). In this way, taking into account that the intervention groups will be carried out in the health care centers of 7 different entities each will have to recruit 24 patients, 12 for each experimental condition.

Data collection: the professional who makes the referral of the patients to the study will be responsible for reviewing fulfillment of the inclusion and exclusion criteria. Patients fulfilling the inclusion criteria will receive an explanation of the study and if they accept to participate, they must provide signed informed consent. The evaluation will be carried out at 3 time points: T0 (basal assessment, prior to initiation of treatment). All the previously described scales will be administered; T1 (post-treatment evaluation), all the scales will be administered and, in addition, the satisfaction perceived with the interventions received will be evaluated; T2 (follow-up evaluation ) at 6 months after completing the intervention all the scales will again be administered. In addition, the number of relapses and hospitalizations during the time interval will be registered. Assessment of the PANSS and GAF should take into account the temporal criterium mentioned in the section of 'Outcomes'. A contingency plan will be considered in the event that difficulties are detected in carrying out any of the phases of the study due to external causes, such as the continuity of the COVID-19 pandemic. This plan will consist of the implementation of interventions and evaluations making use of new technologies. All the centers already have the adequate infrastructure to carry out the project under these conditions.

Data analysis: Firstly, the two groups will be compared with the aim of verifying that there are no significant differences at baseline to confirm that they are comparable after randomization. Comparisons of means for independent samples will be carried out using the Student's t-test for continuous variables and the Chi-square test for categorical variables. The variables of the principal analysis will be the difference between the scores of the two groups (REHACOP+MCT and MCT) in the scores of the scales assessing clinical and personal/psychological recovery. The secondary results will be the differences in other assessments of social functioning, cognitive biases, and social cognition on comparing the two experimental conditions. Changes in the scores of these scales will be analyzed using regression methods for repeated measures, with the post-treatment score of the scales as the dependent variable and the basal score and the REHACOP+MCT group as the co-variables. Temporal stability of the results at 6 months will be assessed using the follow-up score as the dependent variable and evaluating how this affects the basal score, post treatment and the experimental condition. The statistical analyses will be performed according to intention to treat (ITT) without imputing the lost values. Gender, antipsychotic medication, and disease evolution time will be considered as control variables.

Limitations:

One of the limitations of this clinical trial might be the loss to follow-up. To compensate for these losses the sample size will be increased by 20%. It is expected that the losses to follow-up will be similar in the two groups. Otherwise, this variable will be considered as an indicator of the acceptability of treatment.

- Ethical considerations: All the people who participate in the trial will sign the informed consent that takes into account the Declaration of Helsinki and the Organic Law 03/2018 of December 5. In the cases of minors informed consent will be signed by the legal guardians The project will be evaluated by each of the Ethics Committees of the participating centers.

Participants will be informed that the data obtained will only be used for purposes related to the investigation and data confidentiality will be guaranteed according to the provisions of Organic Law 03/2018, of December 5 and Regulation (EU) 2016/679 of the European Parliament and of the Council, of April 27, 2016 and data protection (RGPD). The data management plan generated by the project, all information will be stored and managed in a secure and confidential manner, in accordance with the provisions of Organic Law 03/2018. In order to scrupulously respect the current legislation, the following measures will be taken:

1. Personal data will be pseudonymized. The identifying data are separated from the variables studied in the study. Therefore, a technical and functional separation will be made between the research team and those who perform the pseudonymization and retain the information that allows the reidentification of the participant. Pseudonymized data will only be accessible to the research team when: i) there is an express commitment to confidentiality and no re-identification activity, and ii) specific security measures are taken to prevent re-identification and access to unauthorized personal.
2. The person receiving the informed consent and custody will be different from the person who will process the data, or if this is not possible, the entire research team will sign an express commitment of confidentiality not to carry out re-identification activities. The signed informed consents will be kept under lock and key and out of the reach of the research team in a generic sense.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one of the e following diagnostics according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5): schizophrenia, schizophreniform disorder, delusional disorder, brief psychotic disorder, schizoaffective disorder, and non specified schizophrenia spectrum disorder and other psychotic disorders.
* Be in a stable clinical phase (without psychiatric hospitalization in the last 3 months).
* Have good adherence to pharmacological treatment.
* T-score < 40 in any cognitive outcome measured by TAVEC, CPT-IP, TMT, Stroop, WSCT, FAS and WAIS (Vocabulary, Digit Forward, Digit Backwards and Digit Symbol Coding.
* Willing to participate in the study expressed by providing signed informed consent.

Exclusion Criteria:

* Presence of traumatic brain lesion, dementia or intellectual discapacity (IQ <70).
* Positive and Negative Syndrome Scale (PANSS) score >= 5 in hostility and lack of cooperation and >= 6 in suspiciousness.
* Presence of an additional diagnosis of severe disorder related to substances.
* Having participated in a CR and/or MCT intervention in the year prior to incorporation into the study.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CLINICAL RECOVERY | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Includes: a) CLINICAL REMISSION: based on the criteria of the Remission in Schizophrenia Working Group (RSWA) of Andreasen et al. (2005), which includes one criterium of severity measured with 7 items of the PANSS scale and one temporal criterium that requires the maintenance of the criterium of severity during 6 months or more; and b) FUNCTIONAL RECOVERY: based on the criteria defined by the German Research Network on Schizophrenia (GRNS group) (Schennach-Wolff et al., 2009), which includes one criterium of severity based on the GAF scale and one temporal criterium of maintaining the criterium of severity during 6 months or more.
FUNCTIONAL RECOVERY | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  To be measured with the STORI test.

SECONDARY OUTCOMES:
Assesment instruments | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  A sociodemographic and clinical questionnaire created by the investigators of this study will be given with the aim of collecting the following data: age, gender, education, civil status, coexistence, current professional situation, total number of psychotic episodes, age at the first episode, substance use, type of treatments received (past and present), duration of untreated psychosis (DUP), relapses, number of hospitalisations, diagnosis according to the DSM-5, referral centre, family history, grade of satisfaction with care received, among others.
Social Cognition. Recognition of emotion | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  The facial emotion recognition test will be used (Baron-Cohen et al., 1997; Huerta-Ramos et al., 2017) constituted by 20 photographs expressing 10 basic and 10 complex emotions.
Social Cognition. Hinting Task (Corcoran et al., 1995; Gil et al., 2012) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Includes different stories for evaluating the interpretation of social situations.
Social Cognition. Internal, Personal and Situational Attributions Questionnaire (IPSAQ) (Kinderman & Bentall, 1996; Diez-Alegría, 2006) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  The IPSAQ has 32 items which describe 16 positive and 16 negative social situations. For each situation the person must decide whether the cause is internal, personal or situational.
Ball task (Dudley et al.,1997). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Jumping to conclusions (JTC) will be evaluated with the ball task. This is a task of probabilities in which the persons have to make a decision as to which box a ball belongs. The task will be used with a probability of 85%-15%, 60%-40% and with emotional tasks. JTC will be considered as making a decision after the extraction of one or two balls (Dudley et al., 2016).
Cognitive Bias Questionnaire (CBQ) (Peters et al., 2013; Gutiérrez-Zotes, in press). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  This questionnaire evaluates themost frequent cognitive biases in psychotic disorders. intentionality, catastrophism, dichotomic thinking, JTC and reasoning based on emotions.
Beck Cognitive Insight Scale (BCIS) (Beck et al., 2004; Guitiérrez-Zotes et al., 2012). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  This is a self applied questionnaire including 15 items which collect information on the capacity to correct erroneous judgements in two subscales: self-reflection and self-certainty.
Social Functioning Scale (SFS) (Birchwood et al., 1990; Torres and Olivares, 2000). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  This scale was designed with the aim of evaluating areas of social functioning that are crucial for persons with schizophrenia to remain in the community.
Cognitive functioning. | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  A battery of neuropsychological tests will be carried out to evaluate the domain of general cognitive functioning (Weschler Intelligence Scale [WAIS] (Weschler, 1999), to estimate the IQ using 4 subtests (vocabulary, similarities, block design and matrix reasoning), and specific domains of cognitive functioning.
Global Assessment Functioning (GAF) (Endicott et al., 1976). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  This scale measures the general functioning of the patient on a scale from 0 to 100, with higher scores indicating better functioning. This scale can offer a score on clinical functioning (GAF-C) and another on social functioning (GAF-S).
Positive and negative syndrome scale (PANSS) (Kay et al., 1987; Peralta and Cuesta, 1995). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  The PANSS evaluates positive and negative symptoms and provides a score of general psychopathology.
Continuous Performance Test II (CPT-II) (Conners, 2000); Trail Making Test (TMT) (Reitan,1993). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Attention
Rey Auditory Verbal Learning Test (RAVLT) (Rey, 1964) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Learning and verbal memory
Wisconsin Card Sorting Test (WCST) (Bergs et al., 1948) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Executive functions
Trail Making Test (TMT-B) (Reitan, 1993) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Executive functions
Stroop Color and Word Test (Stroop, 1935) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Executive functions
Trail Making Test (TMT-A) (Reintan, 1993) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Processing Speed
Controlled Oral Word Association Test (COWAT) (Benton&Hamsher, 1976) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Processing Speed
Letter-number sequencing (Wechsler Adult Intelligence Scale [WAIS]) (Weschler, 1999) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Processing Speed
The Stages of Recovery Instrument (STORI) (Andresen et al., 2006; Lemos et al., 2015) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Will be used to assess 4 components (search and maintain hope, reestablishment of positive identity, find the meaning of life and assume responsibility of one's own life) and 5 stages of the recovery process (moratorium, awareness, preparation, rebuilding and growth). This instrument is made up of 50 items which score in the Likert type scale from 0 to 5. The resulting scores represent the 5 phases of personal/psychological recovery. The scale showing the highest score indicates the stage of recovery in which the patient is at that time.
WHO Quality of Life-BREF 26. (WHOQOL-BREF) (Üstun et al., 1988; Vázquez-Barquero et al., 2000). | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Quality of life
World Health Organization Disability Assessment Schedule (WHO-DAS-II) (Üstun et al., 1988; Vázquez-Barquero et al., 2000) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  It's an instrument designed to assess functioning and disability in six main domains: cognition, mobility, self-care, interpersonal relationships, activities of daily living, and participation in society.
Internalized Stigma of Mental Illness Scale (ISMI) (Ritsher, Otilingama, Grajalesa, 2003) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Stigma
Rosenberg self-esteem scale (RSES) (Rosenberg et al., 1965; Atienza, Balaguer & Moreno, 2000) | It will be administered 1 time before de treatment, 1 time after finishing the treatment and 1 time after 6 months completing the intervention.
  Self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Ana Barajas Velez, Principal Investigator — Universitat Autonoma de Barcelona
Locations (1):
- Universitat Autonoma de Barcelona, Cerdanyola del Vallès, Barcelona, Spain